CLINICAL TRIAL: NCT04403867
Title: The Role of Micrometastasis and Isolated Tumor Cells (ITCs) in Uterine Cancers (Endometrial/Cervical) Submitted to Sentinel Lymph Nodes (SLN) Procedure: an Observational Study
Brief Title: The Role of Micrometastasis and Isolated Tumor Cells (ITCs) in Endometrial and Cervical Cancer. A Multicenter Study.
Acronym: ITCMicroUtCa
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Fabio Martinelli, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT 135/19
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Cancer; Cervical Cancer; Sentinel Lymph Node; Micrometastasis; Sentinel Lymph Node Biopsy; Endometrium Tumor; Endometrial Neoplasms; Cervical Neoplasm; Cervical Tumor; Lymph Node Metastases; Lymph Node Disease
Keywords: endometrial cancer; cervical cancer; sentinel lymph node; low volume disease; survival; recurrence rate; adjuvant therapy; micrometastases; isolated tumor cell; macrometastases; ultrastaging; one-step nucleic acid amplification (OSNA)
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Neoplasm Micrometastasis; Lymphatic Metastasis | interventions — sarcolipin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometrial cancer patients: Patients submitted to Sentinel Lymph Node (SLN) procedure. Patients with lymph nodal disease (macrometastasis, micrometastasis, isolated tumor cells).
  Interventions: Procedure: Sentinel lymph node (SLN) biosy +/- lymphadenectomy
- Cervical cancer patients: Patients submitted to Sentinel Lymph Node (SLN) procedure. Patients with lymph nodal disease (macrometastasis, micrometastasis, isolated tumor cells).
  Interventions: Procedure: Sentinel lymph node (SLN) biosy +/- lymphadenectomy

INTERVENTIONS:
Procedure: Sentinel lymph node (SLN) biosy +/- lymphadenectomy — Evaluation of type and volume of lymph nodal disease
  Other Names: Pathological evaluation of lymph nodes (standard H&H + ultrastaging or OSNA)

SUMMARY:
The role of small-volume lymph node disease (ITC and micro metastases) among patients with endometrial or cervical cancer submitted to sentinel node (SLN) procedure is not clearly defined.

This study was designed to create a dataset of patients with lymph nodal disease. Data on type and volume of lymph nodal disease, therapeutic choices and oncological outcomes (DFS, OS, recurrence rate) will be collected and analyzed.

This will allow to define the groups of patients who may need or for whom it can be avoided any adjuvant treatment on the basis of lymph node status.

ELIGIBILITY:
Inclusion Criteria:

* Early stage endometrial cancer scheduled for SLN procedure
* Early stage cervical cancer scheduled for SLN procedure
* Pathological evaluation of SLNs with standard ultra-staging or one-step nucleic acid amplification (OSNA) for the detection of metastasis
* Presence of lymph nodes metastasis (macrometastasis or low volume disease [micrometastasis and isolated tumor cells])

Exclusion Criteria:

* Previous (<5 years) or concomitant malignancy other than non-melanoma skin cancer
* Advanced/metastatic endometrial cancer
* Locally advanced/metastatic cervical cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with early stage uterine (endometrial or cervical) cancer, who underwent a sentinel lymph node (SLN) procedure with an identification of lymph nodes metastasis (macrometastasis or low volume disease [micrometastasis and isolated tumor cells])
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Survival (Disease free survival [DFS], overall survival [OS]) | through study completion, an average of 3 years
  Evaluation of survival outcomes according to the type and volume of lymph nodal disease
Recurrence rate | through study completion, an average of 3 year
  Evaluation of incidence of recurrences (number of patients having a recurrence) according to the type and volume of lymph nodal disease

SECONDARY OUTCOMES:
Usage of adjuvant therapy in case of small-volume lymph node disease | through study completion, an average of 6 months
  Evaluation of the number of patients receiving or not receiving an adjuvant treatment (radiation therapy, chemotherapy, combinations of the two) in case of small-volume lymph node disease (ITC and micro metastasis)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Martinelli, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Result] Gomez-Hidalgo NR, Ramirez PT, Ngo B, Perez-Hoyos S, Coreas N, Sanchez-Iglesias JL, Cabrera S, Franco S, Benavente AP, Gil-Moreno A. Oncologic impact of micrometastases or isolated tumor cells in sentinel lymph nodes of patients with endometrial cancer: a meta-analysis. Clin Transl Oncol. 2020 Aug;22(8):1272-1279. doi: 10.1007/s12094-019-02249-x. Epub 2019 Dec 20. PMID 31863354
- [Result] Ignatov A, Lebius C, Ignatov T, Ivros S, Knueppel R, Papathemelis T, Ortmann O, Eggemann H. Lymph node micrometastases and outcome of endometrial cancer. Gynecol Oncol. 2019 Sep;154(3):475-479. doi: 10.1016/j.ygyno.2019.07.018. Epub 2019 Jul 22. PMID 31345606
- [Result] Piedimonte S, Richer L, Souhami L, Arseneau J, Fu L, Gilbert L, Alfieri J, Jardon K, Zeng XZ. Clinical significance of isolated tumor cells and micrometastasis in low-grade, stage I endometrial cancer. J Surg Oncol. 2018 Dec;118(7):1194-1198. doi: 10.1002/jso.25259. Epub 2018 Oct 24. PMID 30353577
- [Result] Plante M, Stanleigh J, Renaud MC, Sebastianelli A, Grondin K, Gregoire J. Isolated tumor cells identified by sentinel lymph node mapping in endometrial cancer: Does adjuvant treatment matter? Gynecol Oncol. 2017 Aug;146(2):240-246. doi: 10.1016/j.ygyno.2017.05.024. Epub 2017 May 31. PMID 28577885
- [Result] Goebel EA, St Laurent JD, Nucci MR, Feltmate CM. Retrospective detection of isolated tumor cells by immunohistochemistry in sentinel lymph node biopsy performed for endometrial carcinoma: is there clinical significance? Int J Gynecol Cancer. 2020 Mar;30(3):291-298. doi: 10.1136/ijgc-2019-000934. Epub 2019 Dec 8. PMID 31818860
- [Result] Aloisi A, Casanova JM, Tseng JH, Seader KA, Nguyen NT, Alektiar KM, Makker V, Chiang S, Soslow RA, Leitao MM Jr, Abu-Rustum NR. Patterns of FIRST recurrence of stage IIIC1 endometrial cancer with no PARAAORTIC nodal assessment. Gynecol Oncol. 2018 Dec;151(3):395-400. doi: 10.1016/j.ygyno.2018.09.021. Epub 2018 Oct 2. PMID 30286945
- [Result] Nica A, Gien LT, Ferguson SE, Covens A. Does small volume metastatic lymph node disease affect long-term prognosis in early cervical cancer? Int J Gynecol Cancer. 2020 Mar;30(3):285-290. doi: 10.1136/ijgc-2019-000928. Epub 2019 Dec 22. PMID 31871114
- [Result] Delomenie M, Bonsang-Kitzis H, Bats AS, Ngo C, Balaya V, Xuan HTN, Koual M, Mathevet P, Lecuru F. The clinical implication of lymph nodes micrometastases and isolated tumor cells in patients with cervical cancer: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2019 Oct;241:71-76. doi: 10.1016/j.ejogrb.2019.08.010. Epub 2019 Aug 19. PMID 31450214
- [Result] Guani B, Dorez M, Magaud L, Buenerd A, Lecuru F, Mathevet P. Impact of micrometastasis or isolated tumor cells on recurrence and survival in patients with early cervical cancer: SENTICOL Trial. Int J Gynecol Cancer. 2019 Mar;29(3):447-452. doi: 10.1136/ijgc-2018-000089. Epub 2019 Jan 4. PMID 30833435
- [Result] Cibula D, Abu-Rustum NR, Dusek L, Zikan M, Zaal A, Sevcik L, Kenter GG, Querleu D, Jach R, Bats AS, Dyduch G, Graf P, Klat J, Lacheta J, Meijer CJ, Mery E, Verheijen R, Zweemer RP. Prognostic significance of low volume sentinel lymph node disease in early-stage cervical cancer. Gynecol Oncol. 2012 Mar;124(3):496-501. doi: 10.1016/j.ygyno.2011.11.037. Epub 2011 Nov 25. PMID 22120175
- [Result] Cibula D, McCluggage WG. Sentinel lymph node (SLN) concept in cervical cancer: Current limitations and unanswered questions. Gynecol Oncol. 2019 Jan;152(1):202-207. doi: 10.1016/j.ygyno.2018.10.007. Epub 2018 Oct 11. PMID 30318103